CLINICAL TRIAL: NCT07311421
Title: Clinical Study of Non-invasive Blood Glucose Detection Technology Based on Raman Spectroscopy
Brief Title: Raman Spectroscopy-Based Non-Invasive Blood Glucose Detection
Acronym: Raman Glucose
Status: Recruiting | Type: Observational
Sponsor: Beijing Shijitan Hospital, Capital Medical University (Other)
Collaborators: Beijing Institute of Technology (Other)
Responsible Party: Sponsor
Other Study IDs: IIT2025-029-002
Record Dates: First submitted 2025-08-27; First posted 2025-12-31 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-08

CONDITIONS: Diabetes
Keywords: Diabetes Management; Raman Spectroscopy; Non-invasive Blood Glucose Detection; Clinical Application
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control group: Fingertip blood to measure blood sugar
- Raman spectroscopy non-invasive blood glucose measurement group: Blood glucose was measured using Raman spectroscopy noninvasive blood glucose measurement
  Interventions: Diagnostic Test: Raman spectroscopy for blood glucose measurement

INTERVENTIONS:
Diagnostic Test: Raman spectroscopy for blood glucose measurement — Raman spectroscopy non-invasive blood glucose measurement group
  Groups: Raman spectroscopy non-invasive blood glucose measurement group

SUMMARY:
Diabetes is a chronic metabolic disease that is widely prevalent globally, with its incidence rate continuously increasing, posing significant challenges to patient health and public health systems. In China, the number of diabetes patients ranks first in the world, with an adult prevalence rate as high as 12.8%. The core of diabetes management is blood glucose control. However, traditional finger-prick blood testing methods are inconvenient and have low patient compliance. In recent years, non-invasive blood glucose detection technologies have become a research hotspot. Among them, optical methods, especially spectroscopy techniques, are considered to have the most application potential due to their non-invasive, convenient, and stable characteristics.

Raman spectroscopy, as an important branch of spectroscopy, has advantages such as non-invasiveness and high specificity, and has been successfully applied to blood glucose detection in laboratory settings. However, its clinical application is still in the exploratory stage. Foreign research has validated its feasibility, and domestic research has also made certain progress, but overall, it is still in its infancy. This study aims to compare the consistency and accuracy of Raman spectroscopy non-invasive blood glucose detection with traditional finger-prick blood glucose detection by comparing the blood glucose values measured by the two methods at the same time point. Additionally, the study will assess the participants' satisfaction and acceptance of the two methods through questionnaires. The results of this study will provide a scientific basis for the clinical application of Raman spectroscopy technology and offer references for the promotion of non-invasive blood glucose detection technologies. This will help advance the development of non-invasive blood glucose detection technologies and improve the treatment compliance and quality of life of diabetes patients.

ELIGIBILITY:
Inclusion Criteria:

Age range: 18-75 years old. Gender: unlimited. Health status: patients with diagnosed diabetes or healthy volunteers. Nail health status: no obvious infection, discoloration, peeling and other lesions of the nail, so as to ensure the accuracy of Raman spectroscopy measurement.

Willing to participate in the study and sign the informed consent.

Exclusion Criteria:

Nail diseases: such as fungal infections, psoriasis, trauma resulting in nail damage or deformity.

The presence of factors that influenced the measurement results: Participants who used nail polish, fake nails, or nail products. Recent use of drugs containing heavy metals (which may affect nail composition) and skin conditions are not appropriate for such tests.

Pregnant or lactating women. People with serious chronic diseases (such as terminal cancer, end-stage renal disease) or mental illness.

Non-cooperation or inability to complete the entire research process, such as refusal or inability to complete Raman spectrum acquisition.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals aged 18-75 years, either healthy or with diabetes, including both males and females, who have signed the informed consent form. There are no requirements regarding race, education level, or economic status.
Sampling Method: Probability Sample
Enrollment: 49 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-06-10 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Blood glucose value | At the single baseline
  Blood glucose value was assessed as a primary outcome measure in this study. It reflects the concentration of glucose in the blood and serves as a critical indicator for evaluating the metabolic status, particularly in the context of diabetes management.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Beijing Shijitan Hospital, Beijing, Beijing Municipality
  - Beijing Shijitan Hospital, Haidian, Beijing Municipality

IPD SHARING:
Plan to Share IPD: No